CLINICAL TRIAL: NCT04546776
Title: Prevalence and Persistence of SARS-CoV-2 in Stool of COVID-19 Positive Subjects
Brief Title: COVID-19 Persistence in Stool
Acronym: CoPS
Status: Completed | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); James Paget University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: QIB05/2020
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV Infection
Keywords: Faeces; Saliva; Whole-genome shotgun sequencing; COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Faecal and saliva sampling: A minimum of 4 and a maximum of 8 sample sets will be asked for over the study period

SUMMARY:
This is a longitudinal study in which participants that have been confirmed by a National Health Service (NHS) swab test as COVID-19 positive will be asked to provide faecal and saliva samples, and complete short health/lifestyle questionnaires at the time of sampling (referred to as a sample set). The number of sample sets collected from any participant will be dependent on how long the SARS-CoV-2 virus persists within the stool. The investigators aim to collect a minimum of 4 and a maximum of 8 sample sets, and will target all COVID-19-positive subjects, with the exception of those severally ill (e.g. in the intensive care unit (ICU)). The investigators aim to recruit a minimum of 100 and up to 200 participants. To obtain the desired numbers, it may be necessary to continue recruitment during any further United Kingdom (UK) COVID-19 infection peaks.

DETAILED DESCRIPTION:
Approaching participants will mainly be performed in two ways:

1. the Norfolk and Norwich University Hospital (NNUH) online booking system for SARS-CoV-2 testing will have a link to the Quadram Institute Bioscience (QIB) study webpage, which will include the Participant Information Sheet (PIS). When the NHS testing service informs individuals of their test results by text message, the QIB study page Uniform Resource Locator (URL) will be added to the end of the text message for COVID-19 'positive' results. In addition, testing service staff will remind the potential participants of the study if they contact individuals by telephone to inform them of positive COVID-19 results from the test-centre swabs. During this call, potential participants will be asked to provide verbal consent for the study team to contact them for arranging a study talk. Potential participants will be able to contact QIB directly to express interest by email or phone, and can contact QIB to request a hard copy of the PIS be posted to them.
2. NNUH staff will approach in-ward patients positive for COVID-19. Should the patients be interested in learning more, a NNUH staff member will provide them with a copy of the PIS and be available to answer any questions the patients may have. Fully informed written consent of hospitalised COVID-19 patients will be performed by an NNUH nurse using the study consent form.

   * Participants recruited from a non-hospital setting will be consented, using the same consent form as hospitalised patients, over the telephone/internet video by members of the study team who have received the QIB consent training.

Signed copies of these forms will be collected along with the first sample set. In both scenarios, each point will be explained and all questions will be answered to ensure that the participant is fully informed.

The investigators will also be asking participants whether they would be willing to consent to their samples being stored at the Norwich Research Park Biorepository, and whether they would consent to being re-contacted by researchers about possible future research for which they may be eligible. These are both optional, i.e. should the patient choose not to consent to either or both, they will still be able to participate in the study.

Following the recruitment of COVID-19 positive participants the investigators will ask for an initial faecal and saliva sample, and request that the participant completes a health/lifestyle questionnaire. If participants show symptoms the investigators will collect a second set of samples after 48h of symptoms disappearance (specifically, a lack of fever), whereas if participants are asymptomatic the investigators will collect the second set of samples after 7 days. For both types of participants, the investigators will then collect 2 more sample sets every 7 days (day 7: set 3, day 14: set 4). Should either sample test positive then the investigators will continue the same 7-day sampling process until both samples are negative for two consecutive sample sets, or they have given a total of eight faecal and saliva samples. At either of these points, whichever is earliest, the participant will have then completed the study

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years
* Those that live or work within a 40-mile radius of Norwich/Norfolk and Norwich University Hospital
* Those who are confirmed COVID-19 positive by an NHS swab test

Exclusion Criteria:

* Those who are admitted to an NHS Intensive Care Unit
* Any person related to, or living with, any member of the study team
* Those who are part of the Line Manager/supervisory structure of the Chief Investigators
* Those who are unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have tested positive for COVID-19, whether isolated at home or admitted to the Norfolk and Norwich University Hospital. Those admitted to the intensive care unit will not be eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Prevalence and persistence of the SARS-CoV-2 virus in the faeces, and change in associated health status | Weekly for a maximum of 8 weeks
  To verify the prevalence and persistence (starting from symptom onset/diagnosis, and up to seven weeks after recovery) of the SARS-CoV-2 virus in the faeces of people diagnosed with COVID-19 infection.

SECONDARY OUTCOMES:
Viral strain-specific prevalence, associated with change in health status | Weekly for a maximum of 8 weeks
  To use whole-genome sequencing (WGS) to type COVID-19 at the strain level to verify whether different viral strains have a different persistence in stool across participants
Biogeographical viral strain identification, associated with change in health status | Weekly for a maximum of 8 weeks
  To use whole-genome sequencing (WGS) to type COVID-19 at the strain level to verify whether the viral strain(s) found in the gastrointestinal tract are identical to those found in the respiratory tract of participants
Create a SARS-CoV-2 biological sample repository | Through study completion, up to two years
  To create a repository of material (faeces and saliva) and associated data that will be used to understand the association between gastrointestinal health and SARS-CoV-2 infection in future research.

CONTACTS AND LOCATIONS:
Overall Officials: Arjan Narbad, BSc, PhD, Principal Investigator — Quadram Institute Bioscience; Ngozi Franslem-Elumogo, MBBS, DTM&H, FRCPath, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK); Andreas Brodbeck, PhD, FRCA, FICM, Principal Investigator — James Paget University Hospital
Locations (3):
- United Kingdom (3):
  - James Paget University Hospital Foundation Trust, Great Yarmouth, Norfolk
  - Quadram Institute Bioscience, Norwich, Norfolk
  - Norfolk and Norwich University Hospital Foundation Trust, Norwich, Norfolk

IPD SHARING:
Plan to Share IPD: No